CLINICAL TRIAL: NCT03842436
Title: Feasibility and Acceptability of Digital Pills to Monitor PrEP Adherence in MSM With Substance Use
Acronym: DigiPrEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Peter R Chai, Emergency Medicine Physician, Fenway Community Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019P000793
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: HIV/AIDS; Substance Use Disorders; Adherence, Medication
Keywords: PrEP; Substance Use Disorder; Digital Pills; Medication Adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Medication Adherence | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Single group pilot demonstration project
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Digital Pills (Experimental): Digital Pills containing Truvada ingested once daily as PrEP
  Interventions: Device: Digital pill; Drug: Truvada

INTERVENTIONS:
Device: Digital pill — Digital pills over encapsulating Truvada
  Other Names: eTectRx ID Cap
Drug: Truvada — Truvada prescribed with digital pills for PrEP

SUMMARY:
This study deploys a novel digital pill with Emtricitabine/Tenofovir (TDF/FTC) among MSM with substance use to monitor PrEP adherence. The investigators will enroll N=15 HIV uninfected MSM with self reported substance use who are on PrEP or initiating PrEP to use digital pills over encapsulating TDF/FTC for 3 months. The investigators will assess the feasibility of using digital pills in this study population as well as understand the acceptability of digital pills for adherence measurement using semi-structured individual interviews. Additionally, the investigators will measure adherence over time, as well as episodes of suboptimal PrEP adherence.

DETAILED DESCRIPTION:
Eligible study participants will be screened and enrolled at Fenway Health (Boston, MA). Participants will complete a quantitative assessment on their history fo substance use, sexual risk and PrEP adherence, and be trained to use the digital pill for 90 days and instructed to take PrEP daily during the course of the study. Participants will return each month for a study visit to assess their use of the technology. At study visit 1 and 3, we will obtain dried blood spots (DBS) to measure drug levels and to confirm adherence detected by the digital pill. The investigators will also obtain drugs of abuse screens from DBS. At the final study visit (3 months), participants will undergo a semi-structured qualitative interview to understand the user response to digital pills.

ELIGIBILITY:
Inclusion Criteria:

1. MSM (cisgender male)
2. Self-reported use of non-alcohol substances of abuse in past 6 months
3. Currently taking PrEP
4. Has qualifying laboratory tests (Cr, hepatitis B immunization, STI testing and syphilis)
5. Age 18 or older

Exclusion Criteria:

1. Does not speak English
2. HIV positive
3. Identifies as transgender
4. Estimated creatinine clearance <60ml/min
5. Active hepatitis B treatment
6. Does not own a smartphone
7. Taking proton pump inhibitors
8. History of Crohn's disease or ulcerative colitis
9. History of bowel surgery, gastric bypass, bowel stricture
10. History of GI malignancy or radiation to abdomen
11. Unable/unwilling to ingest digital pill

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fenway Health, Boylston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chai PR, Goodman GR, Bronzi O, Gonzales G, Baez A, Bustamante MJ, Najarro J, Mohamed Y, Sullivan MC, Mayer KH, Boyer EW, O'Cleirigh C, Rosen RK. Real-World User Experiences with a Digital Pill System to Measure PrEP Adherence: Perspectives from MSM with Substance Use. AIDS Behav. 2022 Jul;26(7):2459-2468. doi: 10.1007/s10461-022-03594-9. Epub 2022 Jan 28. PMID 35089449
- [Derived] Chai PR, Mohamed Y, Bustamante MJ, Goodman GR, Najarro J, Castillo-Mancilla J, Baez A, Bronzi O, Sullivan MC, Pereira LM, Baumgartner SL, Carnes TC, Mayer KH, Rosen RK, Boyer EW, O'Cleirigh C. DigiPrEP: A Pilot Trial to Evaluate the Feasibility, Acceptability, and Accuracy of a Digital Pill System to Measure PrEP Adherence in Men Who Have Sex With Men Who Use Substances. J Acquir Immune Defic Syndr. 2022 Feb 1;89(2):e5-e15. doi: 10.1097/QAI.0000000000002854. PMID 34753871

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Digital Pills
Started | 16
Completed | 15
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Digital Pills
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: One participant was lost to follow-up.
  years | 32 [29 to 35.5]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant was lost to follow-up.
  Participants
    Female | 0
    Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant was lost to follow-up.
  Participants
    Hispanic or Latino | 4
    Not Hispanic or Latino | 11
    Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One participant was lost to follow-up.
  Participants
    Race: White | 10
    Race: Black / African American | 1
    Race: Asian | 1
    Race: More than one race | 2
    Race: Other | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: One participant was lost to follow-up.
  Participants
    United States | 15
Education [Count of Participants; unit: Participants] — Population: One participant was lost to follow-up.
  Participants
    Some college | 2
    College degree | 7
    Graduate degree/professional | 6
Sexual Orientation [Count of Participants; unit: Participants] — Population: One participant was lost to follow-up.
  Participants
    Homosexual or gay | 13
    Bisexual | 2
STI in prior 12 month [Count of Participants; unit: Participants] — Population: One participant was lost to follow-up.
  Participants
    Yes | 10
    No | 5
Reported substance use [Count of Participants; unit: Participants] — Population: One participant was lost to follow-up.
  Participants
    Alcohol | 14
    Marijuana | 10
    Stimulants | 7
    Hallucinogens | 4
    Other (poppers, amyl nitrate) | 7
Prescribed PrEP [Count of Participants; unit: Participants] — Population: One participant lost to follow-up.
  Participants
    Yes | 14
    No | 1
Nonadherent to PrEP in prior 2 weeks (self-report) [Count of Participants; unit: Participants] — Defined as missing >2 doses of PrEP over the past two weeks. Population: One participant was lost to follow-up. Additionally, the denominator for this variable is 14, as 14 participants had already been prescribed PrEP, and one had not.
  Participants
    number analyzed (Participants) | 14
    Yes | 3
    No | 11

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Digital Pills to Measure PrEP Adherence
Description: Participants' engagement with the digital pill system (DPS) was measured over the 90-day study period. The percentages for the total expected ingestions recorded by DPS each month were compared.
Time Frame: Months 1, 2, and 3
Population: One participant was temporarily lost to follow-up, so they were excluded from analysis.
  In Month 1, the total number of DPS-recorded ingestion events (411) exceeded the total expected ingestion events from pill counts (402), as a result of one participant returning nine more unused pills than anticipated at the end of the month. The total expected ingestions for Month 1 is listed as 411 in the table below for clarity.
Measure: Count of Units; unit: Expected ingestions per pill counts
Units Other Than Participants: Expected ingestions per pill counts
Arm/Group | Digital Pills
Number analyzed (Participants) | 14
Number analyzed (Expected ingestions per pill counts) | 1192
Expected ingestions per pill counts
  Month 1: Total ingestions recorded by DPS: number analyzed (Expected ingestions per pill counts) | 411
  Month 1: Total ingestions recorded by DPS | 411
  Month 2: Total ingestions recorded by DPS: number analyzed (Expected ingestions per pill counts) | 421
  Month 2: Total ingestions recorded by DPS | 368
  Month 3: Total ingestions recorded by DPS: number analyzed (Expected ingestions per pill counts) | 369
  Month 3: Total ingestions recorded by DPS | 320

2. Secondary Outcome: Digital Pill Performance - Number of Recorded Ingestions
Description: The total number recorded ingestions recorded by the digital pill system (DPS) - which included both the number of Reader-detected and manually-reported ingestions - was collected. The Reader-detected ingestions count was used to reflect the number of times the DPS was operated correctly. Successful DPS operation was defined as ingestion of a digital pill, proper use of the wearable Reader, and confirmation of the ingestion on both the Reader and the app. Cumulative data collected at months 1, 2, and 3 are reported in the data table below.
Time Frame: Months 1, 2, and 3
Population: One participant was temporarily lost to follow-up.
Measure: Count of Units; unit: Recorded ingestions
Units Other Than Participants: Recorded ingestions
Arm/Group | Digital Pills
Number analyzed (Participants) | 14
Number analyzed (Recorded ingestions) | 1099
Recorded ingestions
  Reader-detected ingestions | 922
  Manually reported ingestions | 177

3. Secondary Outcome: Digital Pill Performance - System Accuracy
Description: Accuracy of the digital pill system (DPS) in measuring PrEP adherence. To analyze the performance of the DPS, the ground truth of PrEP ingestion events was defined as the pill counts obtained each month (i.e., the number of unused pills returned, subtracted from the number of pills previously dispensed). The number of DPS-recorded ingestions - which included the number of both Reader-detected and manually-reported ingestions - was compared with the aggregate pill count at each monthly timepoint; this was defined as the overall performance metric for the DPS. Cumulative data collected at months 1, 2, and 3 are reported in the data table below.
Time Frame: Months 1, 2, and 3
Population: One participant was temporarily lost to follow-up, so they were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of ingestions DPS recorded
Units Other Than Participants: Expected ingestions based on pill counts
Arm/Group | Digital Pills
Number analyzed (Participants) | 14
Number analyzed (Expected ingestions based on pill counts) | 1192
percentage of ingestions DPS recorded | 92 [91 to 94]

4. Secondary Outcome: Digital Pill Performance - Manually Reported Ingestions
Description: The total number of manually reported ingestions was collected. The percentages for instances of manually reported ingestions were calculated. The two instances for manually recording ingestions included, a lack of engagement with the Reader or failure to use the Reader properly, and when reported ingestion was not detected by the Reader despite supporting use metrics indicating proper Reader use. Cumulative data collected at months 1, 2, and 3 are reported in the data table below.
Time Frame: Months 1, 2, and 3
Population: One participant was temporarily lost to follow-up.
Measure: Count of Units; unit: Manually-reported ingestions
Units Other Than Participants: Manually-reported ingestions
Arm/Group | Digital Pills
Number analyzed (Participants) | 14
Number analyzed (Manually-reported ingestions) | 177
Manually-reported ingestions
  Lack of engagement with the Reader or failure to use Reader properly | 158
  Instances where reported ingestion was not detected by the Reader despite proper Reader use | 19

5. Secondary Outcome: Digital Pill Performance - Successful Operation of System
Description: The total number of instances in which ingestions were successfully detected by the Reader (i.e., the radio frequency emitter was activated, and the ingestion was recorded by the DPS) was collected. The total number of instances in which manually reported ingestions were not detected by the Reader, despite supporting use metrics (e.g., accelerometer data) indicating proper Reader use was also collected. These counts were combined and interpreted as the number of times that the DPS was operated correctly. Cumulative data collected at months 1, 2, and 3 are reported in the data table below.
Time Frame: Months 1, 2, and 3
Population: One participant was temporarily lost to follow-up.
Measure: Count of Units; unit: Ingestions successfully detected by DPS
Units Other Than Participants: Ingestions successfully detected by DPS
Arm/Group | Digital Pills
Number analyzed (Participants) | 14
Number analyzed (Ingestions successfully detected by DPS) | 941
Ingestions successfully detected by DPS
  Reader-detected digital pill ingestions that activated radio frequency emitter | 922
  Manually reported digital pill ingestions with supporting use metrics indicating proper Reader use | 19

6. Secondary Outcome: Dried Blood Spot Correlation With Digital Pill Adherence
Description: We dichotomized TFV-DP levels using a cutoff of ≥700 fmol/punch to indicate at least four doses of PrEP ingested per week. Using TFV-DP in DBS <700 vs ≥700 fmol/punch as a dichotomous variable, and considering the granular continuous adherence data from the digital pill, we then calculated a point biserial correlation between TFV-DP in DBS and digital pill adherence. Additionally, drug concentrations of tenofovir diphosphate as measured in dried blood spot collection at months one and three were compared to DPS-recorded PrEP adherence.
Time Frame: Months 1 and 3
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Units Other Than Participants: Paired DBS samples
Arm/Group | Digital Pills
Number analyzed (Participants) | 15
Number analyzed (Paired DBS samples) | 22
correlation coefficient
  Point-biserial correlation | 0.58 [0.21 to 0.80]
  Pearson's correlation for month one | 0.85 [0.57 to 0.95]
  Pearson's correlation for month three | 0.75 [0.17 to 0.94]

7. Other Pre Specified Outcome: Number of Participants That Completed Qualitative Interview to Evaluate Acceptability of Digital Pills
Description: Acceptability was assessed via individual, semi-structured, qualitative exit interviews conducted at the end of the 90-day study period. The qualitative interview guide was grounded in the Technology Acceptance Model. Questions explored participants' experiences using the digital pill system (DPS), including facilitators and barriers to use, engagement with the technology, and willingness to use the DPS long-term.
Time Frame: Month 3
Population: Qualitative user experience data were collected via interviews from the 15 participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Pills
Number analyzed (Participants) | 15
Participants | 15

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Digital Pills
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
(1) Most participants were White and well-educated, limiting generalizability. (2) Opportunities for technical DPS improvements arose during the study, which required some participants to temporarily manually record doses. (3) The assay utilized for TFV-DP has not been cross-validated and may result in errors in assayed concentration of TFV-DP. (4) Reliance on pill counts may have decreased the measured accuracy of the DPS among participants who did not return unused pills each month.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT03842436/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT03842436/SAP_001.pdf